CLINICAL TRIAL: NCT05872867
Title: An Open-label, Dose-escalation, Phase 1 Study to Investigate the Safety and Tolerability of WM-A1-3389, in Combination With Pembrolizumab in Patients With Advanced or Metastatic Solid Tumors and Non-Small Cell Lung Cancer
Brief Title: Study of WM-A1-3389 in Participants With Advanced or Metastatic Solid Tumors and Non-Small Cell Lung Cancer (MK-3475-E90/KEYNOTE-E90)
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Wellmarker Bio (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: WMA13389-101; MK-3475-E90 (Other: Merck Sharp & Dohme LLC); KEYNOTE-E90 (Other: Merck Sharp & Dohme LLC)
Record Dates: First submitted 2023-04-19; First posted 2023-05-24 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2023-10

CONDITIONS: Advanced Solid Tumor; Metastatic Solid Tumor; Lung Cancer; Colorectal Cancer; Pancreatic Cancer; Cholangiocarcinoma; Head and Neck Cancer; Non Small Cell Lung Cancer
MeSH Terms: conditions — Neoplasm Metastasis; Lung Neoplasms; Colorectal Neoplasms; Pancreatic Neoplasms; Cholangiocarcinoma; Head and Neck Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dose escalation (Stage 1) (Experimental): WM-A1-3389 administered intravenously, weekly for 21 days of each cycle
  Interventions: Biological: WM-A1-3389
- Dose escalation (Stage 2) (Experimental): WM-A1-3389 administered intravenously, weekly for 21 days of each cycle Pembrolizumab 200 mg administered intravenously, every 3 weeks for 21 days of each cycle
  Interventions: Biological: WM-A1-3389; Biological: Pembrolizumab

INTERVENTIONS:
Biological: WM-A1-3389 — Anti-IGSF1 (Immunoglobulin superfamily member 1)
Biological: Pembrolizumab — Anti-PD-1(Programmed cell death protein 1)
  Other Names: KEYTRUDA®
  Arms: Dose escalation (Stage 2)

SUMMARY:
The purpose of the present study is to determine the safety, tolerability, and efficacy of WM-A1-3389 in combination with pembrolizumab in participants with advanced or metastatic solid tumors and non-small cell lung cancer (NSCLC).

ELIGIBILITY:
Inclusion Criteria:

[Stage 1: monotherapy]

1. Be ≥19 and <75 years of age
2. Participant with histologically and/or cytologically confirmed diagnosis of unresectable advanced or metastatic solid tumors that have been confirmed as progressed disease after standard of care or for which no further standard therapy is available due to intolerance or incompatibility
3. IGSF1 positive expression
4. Have measurable disease defined as at least one lesion based on Response Evaluation Criteria In Solid Tumors (RECIST) v1.1
5. Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
6. Have life expectancy ≥ 12 weeks
7. Have adequate organ functions defined as the following laboratory test criteria at screening (During the screening phase, one re-test will be permitted):

   1. Absolute neutrophil count (ANC) ≥ 1,500/mm3
   2. Platelet count ≥ 100,000/mm3
   3. Hemoglobin (Hb) ≥ 9 g/dL
   4. Total bilirubin ≤ 1.5 X Institutional Upper Limit of Normal (IULN) (Not applicable to patients with Gilbert syndrome)
   5. Serum creatinine ≤ 1.5 X IULN
   6. Aspartate aminotransferase (AST) and/or Alanine aminotransferase (ALT) ≤ 2.5 X IULN (AST and ALT ≤ 5 X IULN in patients with confirmed liver metastasis)
   7. Prothrombin time (PT) ≤ 1.5 X IULN *IULN: Institutional Upper Limit of Normal
8. Have provided archival tumor tissue sample obtained within 3 months prior to IP administration or newly obtained biopsy
9. Have agreed to undergo up to 2 tumor tissue biopsies after IP administration
10. Participant (or legally acceptable representative if applicable) provides written informed consent for the trial

[Stage 2: Combination therapy]

1. Be ≥ 19 and < 75 years of age
2. Participant with histologically and/or cytologically confirmed diagnosis of unresectable advanced or metastatic NSCLC

   1. Have been confirmed as progressive disease after standard of care or for which no further standard therapy is available due to intolerance or incompatibility
   2. Have been confirmed as progressive disease during or after anti-cancer therapy including programmed cell death protein 1 (PD-1) inhibitors and programmed cell death-Ligand 1 (PD-L1) inhibitors
   3. IGSF1 positive expression
   4. PD-L1 low or negative expression (tumor proportion score [TPS] < 50%)
3. Have measurable disease defined as at least one lesion based on Response Evaluation Criteria In Solid Tumors (RECIST) v1.1
4. Have ECOG performance status score of 0 or 1
5. Have life expectancy ≥ 12 weeks
6. Have adequate organ functions defined as the following laboratory test criteria at screening (During the screening period, one re-test will be permitted):

   1. Absolute neutrophil count (ANC) ≥ 1500/mm3
   2. Platelet count ≥ 100,000/mm3
   3. Hemoglobin (Hb) ≥ 9 g/dL
   4. Total bilirubin ≤ 1.5 X IULN (Not applicable to patients with Gilbert's syndrome)
   5. Serum creatinine ≤ 1.5 X IULN
   6. Aspartate aminotransferase (AST) or Alanine aminotransferase (ALT) ≤ 2.5 X IULN (AST and ALT ≤ 5 X IULN in patients with confirmed liver metastasis)
   7. Prothrombin time (PT) ≤ 1.5 X IULN *IULN: Institutional Upper Limit of Normal
7. Have provided archival tumor sample obtained within 3 months prior to IP administration or newly obtained biopsy prior to IP administration
8. Have agreed to undergo up to 2 tumor tissue biopsies after IP administration
9. Participant (or legally acceptable representative if applicable) provides written infromed consent for the trial

Exclusion Criteria:

[Common]

1. Have experienced hypersensitivity to IP, any of its excipients or other monoclonal antibody
2. Have any of the following documented medical history or surgical/procedure history:

   1. Other primary malignant tumor (subject may be enrolled if they have neither received any treatment nor experienced disease progression within 3 years) or hematologic malignancy
   2. Major surgery within 4 weeks or minor surgery within 2 weeks prior to IP administration
   3. Clinically significant arrhythmia, acute myocardial infarction, unstable angina pectoris, or New York Heart Association (NYHA) class Ⅲ or Ⅳ heart failure within 6 months prior to IP administration
   4. Severe cerebrovascular disease within 6 months prior to IP administration
   5. Pulmonary thrombosis, deep vein thrombosis, bronchial asthma, obstructive pulmonary disease, or other severe or life-threatening lung diseases (e.g., acute respiratory distress syndrome, lung failure) considered to be inappropriate for study participationt, within 6 months prior to IP administration
   6. Pneumonia or interstitial lung disease requiring steroids

   f. Infection requiring systemic antibiotics or antiviral agents, etc. or uncontorlled Grade ≥ 3 active infectious diseases within 2 weeks prior to IP administration g. Risk factors of ileus or intestinal perforation (including but not limited to history of acute diverticulitis, intra-abdominal abscess, and abdominal carcinomatosis) h. Auto-immune diseases
3. Have any of the following diseases:

   1. Central nervous system or brain metastasis that is uncontrolled or with clinically significant symptoms (except for patients who stopped systemic corticosteroids at least 4 weeks before IP administration and have been stable for at least 4 weeks)
   2. Abnormal ECG regarded as clinically significant by the investigator
   3. Uncontrolled hypertension (systolic blood pressure [SBP] > 160 mmHg or diastolic blood pressure [DBP] > 100 mmHg)
   4. Active infection requiring treatment
   5. Active hepatitis B or C virus infection
   6. History of human immunodeficiency virus infection (HIV) infection
   7. Symptomatic ascites or pleural effusion (except for patients who were treated and clinically stable)
   8. Diseases that may affect the study results based on the judgement of the investigator
4. Have any of the following medication or treatment history:

   1. Anticancer therapy (chemotherapy, hormonal therapy, targeted therapy, or radiotherapy) within 4 weeks prior to IP administration
   2. Immunotherapy such as anti-PD-1, anti PD-L1, anti-cytotoxic T-lymphocyte-associated protein 4 (CTLA-4), etc. within 4 weeks prior to IP administration
   3. Treatment with live attenuated vaccine within 4 weeks prior to IP administration
   4. Treatment with drugs classified as Immunosuppressants, immunomodulators, or immunocytokines within 1 week prior to IP administration (Immunosuppressants, topical corticosteroids, prednisolone 10 mg/day or ≤ equivalent dose of systemic corticosteroids may be permitted for the treatment or prevention of AEs.)
   5. Allogeneic bone marrow or solid organ transplantation
5. Pregnant women, lactating women or men/women of child-bearing potential who are unwilling to maintain abstinence or use adequate methods of contraception or do not consent to refrain from donation of sperm/ova for at least 6 months after the last IP administration

   * Adequate methods of contraception
   1. Oral or injectable hormonal therapy
   2. Implantation of intrauterine device or intrauterine system
   3. Surgical sterilization (vasectomy, tubal ligation, etc.)
6. Have received any other IP or implantation of investigational medical device within 4 weeks prior to IP administration in the present study
7. Patients who are considered ineligible or unable to participate in the study for other reasons based on the judgement of the investigator

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2024-03-14 (Estimated); Primary Completion 2026-02-22 (Estimated); Study Completion 2026-02-22 (Estimated)

PRIMARY OUTCOMES:
Incidence of Dose Limit Toxicities (DLT) | At the end of Cycle 1 (each cycle is 21 days)
Number of Participants Who Experienced an Adverse Event (AE) | Up to 6 Cycles (18 weeks)
Frequency of dose discontinuation and dose reduction due to ADRs | Up to 6 Cycles (18 weeks)

SECONDARY OUTCOMES:
Objective response rate (ORR) based on Response Evaluation Criteria in Solid Tumor (RECIST) v1.1 | Screening, Subsequent Cycles (every 6 weeks), EOT (up to 18 weeks)
Disease control rate (DCR) based on RECIST v1.1 | Screening, Subsequent Cycles (every 6 weeks), EOT (up to 18 weeks)
Disease control rate (DCR) based on Immune RECIST (iRECIST) | Screening, Subsequent Cycles (every 6 weeks), EOT (up to 18 weeks)
Duration of response (DOR) based on RECIST v1.1 | Screening, Subsequent Cycles (every 6 weeks), EOT (up to 18 weeks)
Duration of response (DOR) based on iRECIST | Screening, Subsequent Cycles (every 6 weeks), EOT (up to 18 weeks)
Overall survival (OS) | every 12 weeks after EOT (18 weeks)
Progression free survival (PFS) based on RECIST v1.1 | Screening, Subsequent Cycles (every 6 weeks), EOT (up to 18 weeks)
Progression free survival (PFS) based on iRECIST | Screening, Subsequent Cycles (every 6 weeks), EOT (up to 18 weeks)
Target tumor size | Screening, Subsequent Cycles (every 6 weeks), EOT (up to 18 weeks)
  Maximum rate of change in the sum of the maximum length of the target lesion For target tumor size, the number of subjects, average, standard deviation, median, minimum, and maximum values by each dosing group are presented.
Time to progression (TTP), time to response (TTR), time to failure (TTF), and other assessable efficacy endpoints | Screening, Subsequent Cycles (every 6 weeks), EOT (up to 18 weeks)
Maximum Concentration (Cmax) of WM-A1-3389 or WM-A1-3389 with Pembrolizumab | Cycle 1, Cycle 2, Subsequent Cycles up to EOT (up to 18 weeks)
Maximum Concentration at steady state (Cmax,ss) of WM-A1-3389 or WM-A1-3389 with Pembrolizumab | Cycle 1, Cycle 2, Subsequent Cycles up to EOT (up to 18 weeks)
Minimum Concentration (Cmin) of WM-A1-3389 or WM-A1-3389 with Pembrolizumab | Cycle 1, Cycle 2, Subsequent Cycles up to EOT (up to 18 weeks)
Minimum Concentration at steady state (Cmin,ss) of WM-A1-3389 or WM-A1-3389 with Pembrolizumab | Cycle 1, Cycle 2, Subsequent Cycles up to EOT (up to 18 weeks)
Average Concentration at steady state (Cav,ss) of WM-A1-3389 or WM-A1-3389 with Pembrolizumab | Cycle 1, Cycle 2, Subsequent Cycles up to EOT (up to 18 weeks)
Area under the curve (AUC) of WM-A1-3389 or WM-A1-3389 with Pembrolizumab | Cycle 1, Cycle 2, Subsequent Cycles up to EOT (up to 18 weeks)
Area under the curve (AUC) from 0 to infinity of WM-A1-3389 or WM-A1-3389 with Pembrolizumab | Cycle 1, Cycle 2, Subsequent Cycles up to EOT (up to 18 weeks)
Time to maximum concentration of WM-A1-3389 or WM-A1-3389 with Pembrolizumab | Cycle 1, Cycle 2, Subsequent Cycles up to EOT (up to 18 weeks)
Time to maximum concentration at steady state of WM-A1-3389 or WM-A1-3389 with Pembrolizumab | Cycle 1, Cycle 2, Subsequent Cycles up to EOT (up to 18 weeks)
Half life of WM-A1-3389 or WM-A1-3389 with Pembrolizumab | Cycle 1, Cycle 2, Subsequent Cycles up to EOT (up to 18 weeks)
Peak trough fluctuation (PTF) of WM-A1-3389 or WM-A1-3389 with Pembrolizumab | Cycle 1, Cycle 2, Subsequent Cycles up to EOT (up to 18 weeks)
Accumulation ratio (AR) of WM-A1-3389 or WM-A1-3389 with Pembrolizumab | Cycle 1, Cycle 2, Subsequent Cycles up to EOT (up to 18 weeks)
Clearance rate (CL) of WM-A1-3389 or WM-A1-3389 with Pembrolizumab | Cycle 1, Cycle 2, Subsequent Cycles up to EOT (up to 18 weeks)
Volume of distribution (Vz) of WM-A1-3389 or WM-A1-3389 with Pembrolizumab | Cycle 1, Cycle 2, Subsequent Cycles up to EOT (up to 18 weeks)
Number of participants with anti-WM-A1-3389 antibodies (Stage 1 only) | Up to EOT (up to 18 weeks)

CONTACTS AND LOCATIONS:
Locations (2):
- South Korea (2):
  - Seoul St. Mary's Hospital, Seoul, Seocho-gu
  - Incheon St. Mary's Hospital, Incheon, Yeonsu-gu